CLINICAL TRIAL: NCT05916950
Title: The THOR IDE Study
Acronym: THOR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Philips Clinical & Medical Affairs Global (Industry)
Collaborators: NAMSA (Other); Syntropic Corelab (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 200201
Record Dates: First submitted 2023-06-07; First posted 2023-06-23 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Peripheral Artery Disease; Peripheral Artery Stenosis; Peripheral Artery Calcification; PAD
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Intervention Model Description: Prospective, single-arm, multicenter, and open-label study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Thor Treatment (Experimental): Treatment with the Thor system
  Interventions: Device: Thor laser atherectomy

INTERVENTIONS:
Device: Thor laser atherectomy — Treatment of de novo calcified lesions with laser atherectomy and calcium modification using the Thor system
  Other Names: Thor calcium modification

SUMMARY:
The goal of this clinical trial is to test the Thor system in adult (≥ 18 year old) patients with de novo (new, never treated) calcified lesions in infrainguinal (leg) arteries (peripheral artery disease or PAD).

The main question[s] it aims to answer are:

* Is the Thor system safe in treating these lesions
* Does the Thor system work to treat these lesions

Participants will:

* Receive treatment with the Thor system
* Have follow-up visits at Discharge, 30 days, 6 months, and 12 months

DETAILED DESCRIPTION:
Up to 30 sites in the U.S. will be selected to do this study.

Patients with pain in their legs when walking and/or resting that is due to lack of blood flow to their legs may be able to join the study. To join the study patients must also have blockages in their leg arteries that meet the study criteria.

Before the Thor procedure, patients will have a screening visit that includes a review of their medical records, questions about their medical history and medications taken for blood thinning or circulation, a physical examination of their legs, a test to check the blood flow in their legs (by checking arm and leg blood pressures), blood tests, and a pregnancy test if they are a female able to have children. Patients will also answer questions about any trouble they have had with walking in the last week and their overall quality of life.

All patients in the study will have treatment with the Thor system. There is no "control group" (a group of patients that receives only standard treatment or receives no treatment at all) in this study. During the procedure, the doctor will take x-ray pictures of the leg arteries. They may also use other treatments such as angioplasty balloons, drug-coated balloons, stents, and filters that collect blood clots, if needed.

Patients treated with the Thor system will be watched until they are ready to go home or up to 24 hours after the procedure if they do not go home right away. Before they go home they will have a test to check the blood flow to their legs (by checking arm and leg blood pressures) and be checked for any adverse events.

Patients will return for visits at 30 days, 6 months, and 12 months after the Thor procedure. At these visits patients will be asked questions about their medical history and medications taken for blood thinning or circulation, have a physical examination of their legs, have a test to check the blood flow in their treated leg (by checking arm and leg blood pressures), have an ultrasound of their treated leg, and be checked for any adverse events. Patients will also answer questions about any trouble they have had with walking in the last week and their overall quality of life.

It will take up to 24 months (2 years) to enroll all of the patients in the study. Patients who join the study will be in the study for about 12 months (1 year) and will have all of the visits with their doctor that they would normally have for their PAD.

ELIGIBILITY:
Inclusion Criteria:

* Patient age is ≥18 years
* Patient agrees to participate and to comply with the protocol by signing an IRB approved patient consent form
* Patient is able to walk unassisted or with non-motorized assistive devices
* Patient has PAD with documented Rutherford Class 2-4 of the target limb
* Anticipated life expectancy >12 months, in the opinion of the investigator at the time of enrollment.

Angiographic Inclusion Criteria:

* Patient has de novo atherosclerotic disease of the native SFA and/or the popliteal arteries
* Target lesion has ≥70% diameter stenosis by investigator via visual assessment
* Target lesion length ≤150mm. Total treatment zone may not exceed 150mm, and may include one or more lesions.
* Chronic total occlusion lesion length is <100mm of the total ≤150mm target lesion
* Minimum reference vessel diameter (RVD) 4.0mm by visual estimate
* Target lesion crossed and intraluminal guidewire placement confirmed; successful crossing defined as tip of the guidewire distal to the target lesion in the absence of flow limiting dissections or perforations
* At least one patent tibial vessel (defined as <50% stenosis) with runoff to the foot
* Target lesion has moderate to severe calcification graded using the Peripheral Academic Research Consortium (PARC) criteria

Exclusion Criteria:

* Patient has active infection requiring antibiotic therapy
* Stenting planned within the target lesion
* Known positive for COVID-19 within the last 2 weeks and actively symptomatic
* Pregnant (positive pregnancy test) or currently breast feeding
* Evidence of Acute Limb Ischemia in the target limb within 7 days prior to procedure
* Cerebrovascular accident (CVA) <60 days prior to procedure
* Myocardial infarction <60 days prior to procedure
* History of unstable coronary artery disease or other uncontrollable comorbidity resulting in hospitalization within the last 60 days prior to baseline screening
* Known contraindication to aspirin, or antiplatelet/anti-coagulant therapies required for procedure/follow-up
* Known allergy to contrast media that cannot adequately be premedicated prior to study procedure
* History of Thrombophilia, Heparin-induced Thrombocytopenia (HIT), or Heparin-induced Thrombotic Thrombocytopenia Syndrome (HITTS)
* Serum creatinine ≥2.5mg/dL (unless dialysis-dependent) tested within 30 days prior to procedure
* Planned lower limb major amputation (above the ankle)
* Other surgical or endovascular procedure in the target limb that occurred within 14 days prior to index procedure or is planned on target limb for within 30 days following index procedure, with the exception of diagnostic angiography
* Currently participating in any investigational device or drug clinical trial that, in the opinion of the investigator, will interfere with the conduct of the current study
* The use of specialty balloons, re-entry or additional atherectomy devices is required for treatment of the target lesion.

Angiographic Exclusion Criteria:

* Subject has significant stenosis (>50% stenosis) or occlusion of inflow tract before target treatment zone (e.g. iliac or common femoral) not successfully treated.
* Subject requires treatment of a peripheral lesion on the ipsilateral limb distal to the target site at the time of the index procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 155 (Estimated)
Dates: Start 2024-10-29 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Freedom from Major Adverse Events (MAEs) | 30 Days
  Defined as freedom from MAEs including all-cause mortality, clinically driven target lesion revascularization (CD-TLR), unplanned target limb major amputation, perforations, flow-limiting dissections, and symptomatic distal embolizations that require an intervention to resolve
Procedural Success | At completion of the procedure
  Defined as residual diameter stenosis ≤50% at the end of the procedure as determined by angiographic core lab

SECONDARY OUTCOMES:
Target lesion patency, 30 days | 30 days
  Defined as freedom from CD-TLR and freedom from ≥50% restenosis as determined by duplex ultrasound (DUS) or angiogram
Target lesion patency, 6 months | 6 months
  Defined as freedom from CD-TLR and freedom from ≥50% restenosis as determined by duplex ultrasound (DUS) or angiogram
Target lesion patency, 12 months | 12 months
  Defined as freedom from CD-TLR and freedom from ≥50% restenosis as determined by duplex ultrasound (DUS) or angiogram
Clinically-driven target lesion revascularization | Through 12 months
  Defined as repeat revascularization procedure of the target lesion if PSVR is ≥2.5 by DUS or if angiography shows a percent diameter stenosis >50% and there are worsening clinical symptoms, worsening Rutherford Clinical Category or ABI that is clearly referable to the target lesion.
Technical success | Peri-procedural
  Defined as the ability to deliver the Thor system and achieve residual diameter stenosis ≤50% after treatment with Thor and prior to adjunctive PTA, as confirmed by independent core laboratory assessments of angiographic images
Frequency of peri-procedural adverse events | Within 24 hours of the procedure
  Defined as frequency of adverse events related to the investigational device (Thor system)
Adjunctive devices used with the Thor system | Peri-procedural
  Defined as the use of other devices including angioplasty balloons, drug coated balloons, bailout stents, embolic filters
Target Limb Ankle-Brachial Index (ABI) change, Discharge | Discharge or up to 24 hours after the procedure
  Defined as the change in blood pressure in the upper limb (arm) and lower limb (leg or toes) at discharge compared to the baseline (Screening) value
Target Limb Ankle-Brachial Index (ABI) change, 30 days | 30 days
  Defined as the change in blood pressure in the upper limb (arm) and lower limb (leg or toes) at 30 days compared to the baseline (Screening) value
Target Limb Ankle-Brachial Index (ABI) change, 6 months | 6 months
  Defined as the change in blood pressure in the upper limb (arm) and lower limb (leg or toes) at 6 months compared to the baseline (Screening) value
Target Limb Ankle-Brachial Index (ABI) change, 12 months | 12 months
  Defined as the change in blood pressure in the upper limb (arm) and lower limb (leg or toes) at 12 months compared to the baseline (Screening) value
Rutherford Classification change, 30 days | 30 days
  Defined as the change in Rutherford classification at 30 days compared to the baseline (Screening) value. Rutherford Classification is a staging system to describe reduced blood flow in the lower limb. Rutherford Classifications values range from the least severe (asymptomatic) which is scored a 0 to the most severe (ulceration or gangrene) which is scored a 6.
Rutherford Classification change, 6 months | 6 months
  Defined as the change in Rutherford classification at 6 months compared to the baseline (Screening) value. Rutherford Classification is a staging system to describe reduced blood flow in the lower limb. Rutherford Classifications values range from the least severe (asymptomatic) which is scored a 0 to the most severe (ulceration or gangrene) which is scored a 6.
Rutherford Classification change, 12 months | 12 months
  Defined as the change in Rutherford classification at 12 months compared to the baseline (Screening) value. Rutherford Classification is a staging system to describe reduced blood flow in the lower limb. Rutherford Classifications values range from the least severe (asymptomatic) which is scored a 0 to the most severe (ulceration or gangrene) which is scored a 6.
Freedom from Major Adverse Events (MAEs) | Through 12 months
  Defined as freedom from MAEs including all-cause mortality, clinically driven target lesion revascularization (CD-TLR), unplanned target limb major amputation, and perforations, flow-limiting dissections, and symptomatic distal embolizations that require an intervention to resolve
Change in Short Form Health Survey (SF-36) score, 30 days | 30 days
  Defined as the change in SF-36 score at 30 days compared to the baseline (Screening) value. The SF-36 is a patient-reported survey of patient health. The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.
Change in Short Form Health Survey (SF-36) score, 6 months | 6 months
  Defined as the change in SF-36 score at 6 months compared to the baseline (Screening) value. The SF-36 is a patient-reported survey of patient health. The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.
Change in Short Form Health Survey (SF-36) score, 12 months | 12 months
  Defined as the change in SF-36 score at 12 months compared to the baseline (Screening) value. The SF-36 is a patient-reported survey of patient health. The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.
Change in Walking Impairment Questionnaire (WIQ) score, 30 days | 30 days
  Defined as the change in WIQ score at 30 days compared to the baseline (Screening) value. The WIQ measures self-reported walking impairment, walking distance, walking speed, and stair-climbing ability. In the WIQ there are 21 questions to rate the degree of difficulty with the walking and stair climbing elements. The response for each question is on a 0 to 4 scale, where 0 represents the inability to walk or climb stairs, and 4 represents no difficulty.
Change in Walking Impairment Questionnaire (WIQ) score, 6 months | 6 months
  Defined as the change in WIQ score at 6 months compared to the baseline (Screening) value. The WIQ measures self-reported walking impairment, walking distance, walking speed, and stair-climbing ability. In the WIQ there are 21 questions to rate the degree of difficulty with the walking and stair climbing elements. The response for each question is on a 0 to 4 scale, where 0 represents the inability to walk or climb stairs, and 4 represents no difficulty.
Change in Walking Impairment Questionnaire (WIQ) score, 12 months | 12 months
  Defined as the change in WIQ score at 12 months compared to the baseline (Screening) value. The WIQ measures self-reported walking impairment, walking distance, walking speed, and stair-climbing ability. In the WIQ there are 21 questions to rate the degree of difficulty with the walking and stair climbing elements. The response for each question is on a 0 to 4 scale, where 0 represents the inability to walk or climb stairs, and 4 represents no difficulty.

CONTACTS AND LOCATIONS:
Overall Officials: Pradeep Nair, MD, Principal Investigator — Cardiovascular Institute of the South (CIS); Elizabeth Genovese, MD, Principal Investigator — University of Pennsylvania
Locations (27):
- United States (27):
  - St. Helena Hospital, St. Helena, California
  - Rocky Mountain Regional VA Medical Center, Aurora, Colorado
  - Manatee Memorial Hospital, Bradenton, Florida
  - Guardian Research Organization, Winter Park, Florida
  - Vascular Institute of the Midwest, Davenport, Iowa
  - Cardiovascular Institute of the South, Houma, Louisiana
  - Cardiovascular Institute of the South, Lafayette, Louisiana
  - The Vascular Care Group, Portland, Maine
  - Southcoast Hospitals/Charlton Memorial Hospital, Fall River, Massachusetts
  - Vascular Breakthroughs, Leominster, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Deborah Heart and Lung Center, Browns Mills, New Jersey
  - Heart and Vascular Institute of Central Jersey, New Brunswick, New Jersey
  - Atlantic Medical Imaging of New jersey, Vineland, New Jersey
  - Mount Sinai Hospital, New York, New York
  - New York Presbyterian Hospital/Columbia University Irving Medical Center, New York, New York
  - Vascular Solutions of North Carolina, Cary, North Carolina
  - Premier Cardiovascular Institute, Fairborn, Ohio
  - Ascension St. John, Bartlesville, Oklahoma
  - UPMC, Mechanicsburg, Pennsylvania
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Lankenau Institute for Medical Research, Wynnewood, Pennsylvania
  - The Miriam Hospital, Providence, Rhode Island
  - Vascular Institute of Chattanooga, Chattanooga, Tennessee
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Baylor, Scott & White, The Heart Hospital, Plano, Texas
  - Sentara Health Research Center, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Norgren L, Hiatt WR, Dormandy JA, Nehler MR, Harris KA, Fowkes FG; TASC II Working Group; Bell K, Caporusso J, Durand-Zaleski I, Komori K, Lammer J, Liapis C, Novo S, Razavi M, Robbs J, Schaper N, Shigematsu H, Sapoval M, White C, White J, Clement D, Creager M, Jaff M, Mohler E 3rd, Rutherford RB, Sheehan P, Sillesen H, Rosenfield K. Inter-Society Consensus for the Management of Peripheral Arterial Disease (TASC II). Eur J Vasc Endovasc Surg. 2007;33 Suppl 1:S1-75. doi: 10.1016/j.ejvs.2006.09.024. Epub 2006 Nov 29. No abstract available. PMID 17140820
- [Background] Hirsch AT, Haskal ZJ, Hertzer NR, Bakal CW, Creager MA, Halperin JL, Hiratzka LF, Murphy WR, Olin JW, Puschett JB, Rosenfield KA, Sacks D, Stanley JC, Taylor LM Jr, White CJ, White J, White RA, Antman EM, Smith SC Jr, Adams CD, Anderson JL, Faxon DP, Fuster V, Gibbons RJ, Hunt SA, Jacobs AK, Nishimura R, Ornato JP, Page RL, Riegel B; American Association for Vascular Surgery; Society for Vascular Surgery; Society for Cardiovascular Angiography and Interventions; Society for Vascular Medicine and Biology; Society of Interventional Radiology; ACC/AHA Task Force on Practice Guidelines Writing Committee to Develop Guidelines for the Management of Patients With Peripheral Arterial Disease; American Association of Cardiovascular and Pulmonary Rehabilitation; National Heart, Lung, and Blood Institute; Society for Vascular Nursing; TransAtlantic Inter-Society Consensus; Vascular Disease Foundation. ACC/AHA 2005 Practice Guidelines for the management of patients with peripheral arterial disease (lower extremity, renal, mesenteric, and abdominal aortic): a collaborative report from the American Association for Vascular Surgery/Society for Vascular Surgery, Society for Cardiovascular Angiography and Interventions, Society for Vascular Medicine and Biology, Society of Interventional Radiology, and the ACC/AHA Task Force on Practice Guidelines (Writing Committee to Develop Guidelines for the Management of Patients With Peripheral Arterial Disease): endorsed by the American Association of Cardiovascular and Pulmonary Rehabilitation; National Heart, Lung, and Blood Institute; Society for Vascular Nursing; TransAtlantic Inter-Society Consensus; and Vascular Disease Foundation. Circulation. 2006 Mar 21;113(11):e463-654. doi: 10.1161/CIRCULATIONAHA.106.174526. No abstract available. PMID 16549646
- [Background] Hirsch AT, Criqui MH, Treat-Jacobson D, Regensteiner JG, Creager MA, Olin JW, Krook SH, Hunninghake DB, Comerota AJ, Walsh ME, McDermott MM, Hiatt WR. Peripheral arterial disease detection, awareness, and treatment in primary care. JAMA. 2001 Sep 19;286(11):1317-24. doi: 10.1001/jama.286.11.1317. PMID 11560536
- [Background] Mueller T, Hinterreiter F, Poelz W, Haltmayer M, Dieplinger B. Mortality rates at 10 years are higher in diabetic than in non-diabetic patients with chronic lower extremity peripheral arterial disease. Vasc Med. 2016 Oct;21(5):445-452. doi: 10.1177/1358863X16643603. Epub 2016 Apr 11. PMID 27067137
- [Background] Caro J, Migliaccio-Walle K, Ishak KJ, Proskorovsky I. The morbidity and mortality following a diagnosis of peripheral arterial disease: long-term follow-up of a large database. BMC Cardiovasc Disord. 2005 Jun 22;5:14. doi: 10.1186/1471-2261-5-14. PMID 15972099
- [Background] Dieter RS, Chu WW, Pacanowski JP Jr, McBride PE, Tanke TE. The significance of lower extremity peripheral arterial disease. Clin Cardiol. 2002 Jan;25(1):3-10. doi: 10.1002/clc.4950250103. PMID 11808837
- [Background] Guez D, Hansberry DR, Gonsalves CF, Eschelman DJ, Parker L, Rao VM, Levin DC. Recent Trends in Endovascular and Surgical Treatment of Peripheral Arterial Disease in the Medicare Population. AJR Am J Roentgenol. 2020 May;214(5):962-966. doi: 10.2214/AJR.19.21967. Epub 2020 Feb 25. PMID 32097027
- [Background] Rocha-Singh KJ, Jaff MR, Crabtree TR, Bloch DA, Ansel G; VIVA Physicians, Inc. Performance goals and endpoint assessments for clinical trials of femoropopliteal bare nitinol stents in patients with symptomatic peripheral arterial disease. Catheter Cardiovasc Interv. 2007 May 1;69(6):910-9. doi: 10.1002/ccd.21104. PMID 17377972
- [Background] Minar E, Pokrajac B, Maca T, Ahmadi R, Fellner C, Mittlbock M, Seitz W, Wolfram R, Potter R. Endovascular brachytherapy for prophylaxis of restenosis after femoropopliteal angioplasty : results of a prospective randomized study. Circulation. 2000 Nov 28;102(22):2694-9. doi: 10.1161/01.cir.102.22.2694. PMID 11094034
- [Background] van der Zaag ES, Legemate DA, Prins MH, Reekers JA, Jacobs MJ. Angioplasty or bypass for superficial femoral artery disease? A randomised controlled trial. Eur J Vasc Endovasc Surg. 2004 Aug;28(2):132-7. doi: 10.1016/j.ejvs.2004.04.003. PMID 15234692
- [Background] Schillinger M, Sabeti S, Loewe C, Dick P, Amighi J, Mlekusch W, Schlager O, Cejna M, Lammer J, Minar E. Balloon angioplasty versus implantation of nitinol stents in the superficial femoral artery. N Engl J Med. 2006 May 4;354(18):1879-88. doi: 10.1056/NEJMoa051303. PMID 16672699
- [Background] Pokrajac B, Potter R, Wolfram RM, Budinsky AC, Kirisits C, Lileg B, Mendel H, Sabeti S, Schmid R, Minar E. Endovascular brachytherapy prevents restenosis after femoropopliteal angioplasty: results of the Vienna-3 randomised multicenter study. Radiother Oncol. 2005 Jan;74(1):3-9. doi: 10.1016/j.radonc.2004.08.015. PMID 15683661
- [Background] Krankenberg H, Schluter M, Steinkamp HJ, Burgelin K, Scheinert D, Schulte KL, Minar E, Peeters P, Bosiers M, Tepe G, Reimers B, Mahler F, Tubler T, Zeller T. Nitinol stent implantation versus percutaneous transluminal angioplasty in superficial femoral artery lesions up to 10 cm in length: the femoral artery stenting trial (FAST). Circulation. 2007 Jul 17;116(3):285-92. doi: 10.1161/CIRCULATIONAHA.107.689141. Epub 2007 Jun 25. PMID 17592075
- [Background] Sabeti S, Schillinger M, Amighi J, Sherif C, Mlekusch W, Ahmadi R, Minar E. Primary patency of femoropopliteal arteries treated with nitinol versus stainless steel self-expanding stents: propensity score-adjusted analysis. Radiology. 2004 Aug;232(2):516-21. doi: 10.1148/radiol.2322031345. PMID 15286322
- [Background] Ferreira M, Lanziotti L, Monteiro M, Abuhadba G, Capotorto LF, Nolte L, Fearnot N. Superficial femoral artery recanalization with self-expanding nitinol stents: long-term follow-up results. Eur J Vasc Endovasc Surg. 2007 Dec;34(6):702-8. doi: 10.1016/j.ejvs.2007.07.025. Epub 2007 Oct 24. PMID 17920306
- [Background] Dosluoglu HH, Cherr GS, Lall P, Harris LM, Dryjski ML. Stenting vs above knee polytetrafluoroethylene bypass for TransAtlantic Inter-Society Consensus-II C and D superficial femoral artery disease. J Vasc Surg. 2008 Nov;48(5):1166-74. doi: 10.1016/j.jvs.2008.06.006. Epub 2008 Aug 9. PMID 18692357
- [Background] Dearing DD, Patel KR, Compoginis JM, Kamel MA, Weaver FA, Katz SG. Primary stenting of the superficial femoral and popliteal artery. J Vasc Surg. 2009 Sep;50(3):542-7. doi: 10.1016/j.jvs.2009.04.019. Epub 2009 Jun 21. PMID 19540706
- [Background] Zeller T, Tiefenbacher C, Steinkamp HJ, Langhoff R, Wittenberg G, Schluter M, Buergelin K, Rastan A, Krumsdorf U, Sixt S, Schulte CL, Tubler T, Krankenberg H. Nitinol stent implantation in TASC A and B superficial femoral artery lesions: the Femoral Artery Conformexx Trial (FACT). J Endovasc Ther. 2008 Aug;15(4):390-8. doi: 10.1583/08-2461.1. PMID 18729564
- [Background] Schlager O, Dick P, Sabeti S, Amighi J, Mlekusch W, Minar E, Schillinger M. Long-segment SFA stenting--the dark sides: in-stent restenosis, clinical deterioration, and stent fractures. J Endovasc Ther. 2005 Dec;12(6):676-84. doi: 10.1583/05-1672.1. PMID 16363897
- [Background] Inoue S, Koyama H, Miyata T, Shigematsu H. Pathogenetic heterogeneity of in-stent lesion formation in human peripheral arterial disease. J Vasc Surg. 2002 Apr;35(4):672-8. doi: 10.1067/mva.2002.122021. PMID 11932661
- [Background] Soor GS, Vukin I, Leong SW, Oreopoulos G, Butany J. Peripheral vascular disease: who gets it and why? A histomorphological analysis of 261 arterial segments from 58 cases. Pathology. 2008 Jun;40(4):385-91. doi: 10.1080/00313020802036764. PMID 18446629
- [Background] Lehto S, Niskanen L, Suhonen M, Ronnemaa T, Laakso M. Medial artery calcification. A neglected harbinger of cardiovascular complications in non-insulin-dependent diabetes mellitus. Arterioscler Thromb Vasc Biol. 1996 Aug;16(8):978-83. doi: 10.1161/01.atv.16.8.978. PMID 8696962
- [Background] Shanahan CM, Cary NR, Salisbury JR, Proudfoot D, Weissberg PL, Edmonds ME. Medial localization of mineralization-regulating proteins in association with Monckeberg's sclerosis: evidence for smooth muscle cell-mediated vascular calcification. Circulation. 1999 Nov 23;100(21):2168-76. doi: 10.1161/01.cir.100.21.2168. PMID 10571976
- [Background] Thompson B, Towler DA. Arterial calcification and bone physiology: role of the bone-vascular axis. Nat Rev Endocrinol. 2012 Sep;8(9):529-43. doi: 10.1038/nrendo.2012.36. Epub 2012 Apr 3. PMID 22473330
- [Background] Rocha-Singh KJ, Zeller T, Jaff MR. Peripheral arterial calcification: prevalence, mechanism, detection, and clinical implications. Catheter Cardiovasc Interv. 2014 May 1;83(6):E212-20. doi: 10.1002/ccd.25387. Epub 2014 Feb 10. PMID 24402839
- [Background] Lanzer P, Boehm M, Sorribas V, Thiriet M, Janzen J, Zeller T, St Hilaire C, Shanahan C. Medial vascular calcification revisited: review and perspectives. Eur Heart J. 2014 Jun 14;35(23):1515-25. doi: 10.1093/eurheartj/ehu163. Epub 2014 Apr 16. PMID 24740885
- [Background] Isner JM, Rosenfield K. Redefining the treatment of peripheral artery disease. Role of percutaneous revascularization. Circulation. 1993 Oct;88(4 Pt 1):1534-57. doi: 10.1161/01.cir.88.4.1534. No abstract available. PMID 8403302
- [Background] Schramm KM, DeWitt PE, Dybul S, Rochon PJ, Patel P, Hieb RA, Rogers RK, Ryu RK, Wolhauer M, Hong K, Trivedi PS. Recent Trends in Clinical Setting and Provider Specialty for Endovascular Peripheral Artery Disease Interventions for the Medicare Population. J Vasc Interv Radiol. 2020 Apr;31(4):614-621.e2. doi: 10.1016/j.jvir.2019.10.025. Epub 2020 Feb 29. PMID 32127322
- [Background] Walker KL, Nolan BW, Columbo JA, Rzucidlo EM, Goodney PP, Walsh DB, Atkinson BJ, Powell RJ. Lesion complexity drives the cost of superficial femoral artery endovascular interventions. J Vasc Surg. 2015 Oct;62(4):998-1002. doi: 10.1016/j.jvs.2015.04.450. Epub 2015 Jul 21. PMID 26206581
- [Background] Capek P, McLean GK, Berkowitz HD. Femoropopliteal angioplasty. Factors influencing long-term success. Circulation. 1991 Feb;83(2 Suppl):I70-80. PMID 1825050
- [Background] Herten M, Torsello GB, Schonefeld E, Stahlhoff S. Critical appraisal of paclitaxel balloon angioplasty for femoral-popliteal arterial disease. Vasc Health Risk Manag. 2016 Aug 29;12:341-56. doi: 10.2147/VHRM.S81122. eCollection 2016. PMID 27621646
- [Background] Brodmann M, Werner M, Holden A, Tepe G, Scheinert D, Schwindt A, Wolf F, Jaff M, Lansky A, Zeller T. Primary outcomes and mechanism of action of intravascular lithotripsy in calcified, femoropopliteal lesions: Results of Disrupt PAD II. Catheter Cardiovasc Interv. 2019 Feb 1;93(2):335-342. doi: 10.1002/ccd.27943. Epub 2018 Nov 25. PMID 30474206
- [Background] Brodmann M, Werner M, Brinton TJ, Illindala U, Lansky A, Jaff MR, Holden A. Safety and Performance of Lithoplasty for Treatment of Calcified Peripheral Artery Lesions. J Am Coll Cardiol. 2017 Aug 15;70(7):908-910. doi: 10.1016/j.jacc.2017.06.022. No abstract available. PMID 28797363
- [Background] Adams G, Soukas PA, Mehrle A, Bertolet B, Armstrong EJ. Intravascular Lithotripsy for Treatment of Calcified Infrapopliteal Lesions: Results from the Disrupt PAD III Observational Study. J Endovasc Ther. 2022 Feb;29(1):76-83. doi: 10.1177/15266028211032953. Epub 2021 Aug 12. PMID 34380334
- [Background] Tepe G, Brodmann M, Werner M, Bachinsky W, Holden A, Zeller T, Mangalmurti S, Nolte-Ernsting C, Bertolet B, Scheinert D, Gray WA; Disrupt PAD III Investigators. Intravascular Lithotripsy for Peripheral Artery Calcification: 30-Day Outcomes From the Randomized Disrupt PAD III Trial. JACC Cardiovasc Interv. 2021 Jun 28;14(12):1352-1361. doi: 10.1016/j.jcin.2021.04.010. PMID 34167675
- [Background] Stavroulakis K, Bisdas T, Torsello G, Tsilimparis N, Damerau S, Argyriou A. Intravascular Lithotripsy and Drug-Coated Balloon Angioplasty for Severely Calcified Femoropopliteal Arterial Disease. J Endovasc Ther. 2023 Feb;30(1):106-113. doi: 10.1177/15266028221075563. Epub 2022 Feb 7. PMID 35130782
- [Background] Radaideh Q, Shammas NW, Shammas WJ, Shammas GA. Shockwave Lithoplasty in Combination With Atherectomy in Treating Severe Calcified Femoropopliteal and Iliac Artery Disease: A Single-Center Experience. Cardiovasc Revasc Med. 2021 Jan;22:66-70. doi: 10.1016/j.carrev.2020.06.015. Epub 2020 Jun 11. PMID 32563711
- [Background] Patel MR, Conte MS, Cutlip DE, Dib N, Geraghty P, Gray W, Hiatt WR, Ho M, Ikeda K, Ikeno F, Jaff MR, Jones WS, Kawahara M, Lookstein RA, Mehran R, Misra S, Norgren L, Olin JW, Povsic TJ, Rosenfield K, Rundback J, Shamoun F, Tcheng J, Tsai TT, Suzuki Y, Vranckx P, Wiechmann BN, White CJ, Yokoi H, Krucoff MW. Evaluation and treatment of patients with lower extremity peripheral artery disease: consensus definitions from Peripheral Academic Research Consortium (PARC). J Am Coll Cardiol. 2015 Mar 10;65(9):931-41. doi: 10.1016/j.jacc.2014.12.036. PMID 25744011
- [Background] Dattilo R, Himmelstein SI, Cuff RF. The COMPLIANCE 360 degrees Trial: a randomized, prospective, multicenter, pilot study comparing acute and long-term results of orbital atherectomy to balloon angioplasty for calcified femoropopliteal disease. J Invasive Cardiol. 2014 Aug;26(8):355-60. PMID 25091093
- [Background] Shammas NW, Chandra P, Brodmann M, Weinstock B, Sedillo G, Cawich I, Micari A, Lee A, Metzger C, Palena LM, Rundback J; EX-PAD-03 Investigators. Acute and 30-Day Safety and Effectiveness Evaluation of Eximo Medical's B-Laser, a Novel Atherectomy Device, in Subjects Affected With Infrainguinal Peripheral Arterial Disease: Results of the EX-PAD-03 Trial. Cardiovasc Revasc Med. 2020 Jan;21(1):86-92. doi: 10.1016/j.carrev.2018.11.022. Epub 2018 Nov 29. PMID 30559030
- [Background] Yamamoto Y, Kawarada O, Ando H, Anzai H, Zen K, Tamura K, Tsukahara K, Tsubakimoto Y, Toma M, Nakamura S, Nakamura H, Hozawa K, Yokoi Y, Yasuda S. Effects of high-speed rotational atherectomy in peripheral artery disease patients with calcified lesions: a retrospective multicenter registry. Cardiovasc Interv Ther. 2020 Oct;35(4):393-397. doi: 10.1007/s12928-020-00643-9. Epub 2020 Feb 28. PMID 32112238
- [Background] Zeller T, Langhoff R, Rocha-Singh KJ, Jaff MR, Blessing E, Amann-Vesti B, Krzanowski M, Peeters P, Scheinert D, Torsello G, Sixt S, Tepe G; DEFINITIVE AR Investigators. Directional Atherectomy Followed by a Paclitaxel-Coated Balloon to Inhibit Restenosis and Maintain Vessel Patency: Twelve-Month Results of the DEFINITIVE AR Study. Circ Cardiovasc Interv. 2017 Sep;10(9):e004848. doi: 10.1161/CIRCINTERVENTIONS.116.004848. PMID 28916599
- [Background] Dave RM, Patlola R, Kollmeyer K, Bunch F, Weinstock BS, Dippel E, Jaff MR, Popma J, Weissman N; CELLO Investigators. Excimer laser recanalization of femoropopliteal lesions and 1-year patency: results of the CELLO registry. J Endovasc Ther. 2009 Dec;16(6):665-75. doi: 10.1583/09-2781.1. PMID 19995111
- [Background] Roberts D, Niazi K, Miller W, Krishnan P, Gammon R, Schreiber T, Shammas NW, Clair D; DEFINITIVE Ca(+)(+) Investigators. Effective endovascular treatment of calcified femoropopliteal disease with directional atherectomy and distal embolic protection: final results of the DEFINITIVE Ca(+)(+) trial. Catheter Cardiovasc Interv. 2014 Aug 1;84(2):236-44. doi: 10.1002/ccd.25384. Epub 2014 Feb 5. PMID 24402764
- [Background] Iida O, Urasawa K, Shibata Y, Yamamoto Y, Ando H, Fujihara M, Nakama T, Miyashita Y, Mori S, Diaz-Cartelle J, Soga Y. Clinical Safety and Efficacy of Rotational Atherectomy in Japanese Patients with Peripheral Arterial Disease Presenting Femoropopliteal Lesions: The J-SUPREME and J-SUPREME II Trials. J Endovasc Ther. 2022 Apr;29(2):240-247. doi: 10.1177/15266028211045700. Epub 2021 Sep 13. PMID 34510954
- [Background] Shammas NW, Lam R, Mustapha J, Ellichman J, Aggarwala G, Rivera E, Niazi K, Balar N. Comparison of orbital atherectomy plus balloon angioplasty vs. balloon angioplasty alone in patients with critical limb ischemia: results of the CALCIUM 360 randomized pilot trial. J Endovasc Ther. 2012 Aug;19(4):480-8. doi: 10.1583/JEVT-12-3815MR.1. PMID 22891826
- [Background] Shammas NW, Shammas GA, Jones-Miller S, Shammas WJ, Bou-Dargham B, Shammas AN, Banerjee S, Rachwan RJ, Daher GE. Long-term outcomes with Jetstream atherectomy with or without drug coated balloons in treating femoropopliteal arteries: A single center experience (JET-SCE). Cardiovasc Revasc Med. 2018 Oct;19(7 Pt A):771-777. doi: 10.1016/j.carrev.2018.02.003. Epub 2018 Feb 9. PMID 30420096
- [Background] Gandini R, Pratesi G, Merolla S, Scaggiante J, Chegai F. A Single-Center Experience With Phoenix Atherectomy System in Patients With Moderate to Heavily Calcified Femoropopliteal Lesions. Cardiovasc Revasc Med. 2020 May;21(5):676-681. doi: 10.1016/j.carrev.2019.08.019. Epub 2019 Aug 23. PMID 31488361
- [Background] Burckenmeyer F, Aschenbach R, Diamantis I, Teichgraber U. Excimer laser atherectomy in complex peripheral artery disease: a prospective European registry. J Cardiovasc Surg (Torino). 2021 Apr;62(2):153-161. doi: 10.23736/S0021-9509.21.11569-1. Epub 2021 Jan 22. PMID 33480520